CLINICAL TRIAL: NCT06793839
Title: Pilot Study : Characterization of Early Brain Injury and Delayed Cerebral Ischemia After Aneurysmal Subarachnoid Hemorrhage by Ultrasound Localization Microscopy (ULM) 3D with an Experimental Medical Device (ESRIR)
Brief Title: 3D Contrast Enhanced Acoustic Perfusion Imaging in Adult After Subarachnoid Hemorrhage
Acronym: ESRIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CHU 23-0184; 2023-A01978-37 (Registry Identifier: ID RCB (ANSM))
Record Dates: First submitted 2024-07-10; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: aneurysmal; subarachnoid; hemorrhage; transcranial; doppler; ultrasonography; vasospasm; localizing; microscopy; delayed; cerebral; ischemia; aneurysm; anterior
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hemorrhage; Ischemia; Aneurysm

STUDY DESIGN:
Intervention Model Description: Single group of 15 patients with subarachnoïd hemorrhage
Masking Description: The investigator and care provider can't see the imaging results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasonography localizing microscopy 3D (Experimental): Enhanced (with Sonovue IV 2,4mL x2) transcranial ultrasonography
  Interventions: Device: Transcranial Enhanced Ultrasonography localizing microscopy

INTERVENTIONS:
Device: Transcranial Enhanced Ultrasonography localizing microscopy — 3 bilateral transcranial enhanced (with Sonovue) ultrasonography per patient to visualize cranial arteries of the anterior circulation of the brain
  Other Names: MARIUS

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) is a devastating form of stroke, with three major complications : early brain injury (EBI), vasospasm and delayed cerebral ischemia (DCI). Those patients are often given care in neurocritical care. Imaging is particularly useful to diagnose these complications. Brain imaging includes CT scan, MRI and arteriography which are not easily available and need an intrahospital transportation. Furthermore, intrahospital transportation of critically ill patients is associated with significant complications Here, investigators try to show that a new non-invasive bedside device, based on 3D enhanced ultrasonography, is able to detect principal arteries of anterior circulation of the brain.

DETAILED DESCRIPTION:
Introduction: Aneurysmal subarachnoid hemorrhage (SAH) is a devastating form of hemorrhagic stroke. Majors complications of aneurysmal SAH include early brain injury (EBI), vasospam and delayed cerebral ischemia (DCI). There are currently only few ways through imaging to diagnose those complication. Transcranial doppler (TCD) is an accessible bedside tool which is efficient, but can only provide indirect evidences. Other brain imaging includes CT scan, MRI and arteriography which are not easily available and are associated with intrahospital transportation of critically ill patients and its morbidity. There are several preclinical evidences that 3D enhanced ultrasonography localizing microscopy could show similar images resolution to angiography while being more accessible.

Materials and methods: this study will include patients with aneurysmal SAH. Aneurysm must be of anterior circulation.The investigators will perform a feasibility research with a new medical device based on ultrasonography localizing microscopy. The standard of care will not be changed, but each patient will also get three bilateral transcranial enhanced (with microbubbles from Sonovue) ultrasonography, one for each period at risk (J0-J2, J4-10, J11-J14). The primary outcome will be the quality of time-intensity curve of the contrast agent, in order to show the quality of signal received. Then, as a secondary outcome, images will be compared to clinical findings. As a pilot study, the investigators plan to include only 15 patients in a monocentric trial.

This device could provide real-time information on blood flow and potential complications such as vasospasm or DCI, allowing for earlier intervention and potentially improving outcomes for SAH patients. Additionally, the bedside nature of this device eliminates the need for intrahospital transportation, reducing the risk of complications associated with moving critically ill patients.

This study aims to assess the feasibility and potential benefits of using 3D enhanced ultrasonography localizing microscopy in the management of aneurysmal SAH. The results of this pilot study could pave the way for larger clinical trials and ultimately lead to improved outcomes for patients with this devastating condition.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in neurologic ICU of the CHU Caen, Normandy, for a subarachnoid hemorrhage of the anterior circulation.
* Usable ultrasound temporal window.
* 18 years old and more.
* Consent of the participant or the trusted person.

Exclusion Criteria:

* non-aneurysmal subarachnoid haemorrhage.
* Contraindication to ultrasound contrast agent Sonovue, including allergies to a compound.
* Uncontrolled systemic hypertension.
* Acute respiratory distress syndrome.
* Pregnancy or breastfeeding mother.
* Vulnerable person with guardianship or curatorship.
* Patient not affiliated to french social security system (Sécurité Sociale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Presence of a time-intensity curve (TIC) of contrast agent / Quality of signal | day 0-2 / day 4-10 / day 11-14
  Mathematical models may be used to estimate blood flow parameters after the administration of microbubble contrast agents. A time-intensity curve (TIC) may be created to reflect the intravascular transit of the contrast agent. TICs reflect the average intensity in a region of interest, measured in absolute intensity units, over time in seconds. Plotting TIC in a given frame allows for quantification of various parameters, including time to peak, peak intensity, area under the curve, wash-in and wash-out time, and mean transit time. Some of these parameters, such as peak intensity and area under the curve, reflect local blood volume in the region of interest, whereas, other parameters (time to peak intensity, wash-in/wash-out time) are more reflective of blood flow.

SECONDARY OUTCOMES:
Agreement between data from 3D ultrasonography localizing miroscopy and clinical parameters of early brain injury, cerebral vasospam and delayed cerebral ischemia | day 0-2 / day 4-10 / day 11-14
  Morphology : Visually compare images from ULM and angiography or vasculary atlas Speed : Each side compared to classical temporal doppler ultrasonography Caliber : Mesure of principal arteries' diameter and compare with angiography Perfusion : Time-intensity curve's parameter of each side
Ability to detect principal arteries of anterior circulation | day 0-2 / day 4-10 / day 11-14
  Questionnary filled by the investigator's and research team with the number and size of correct identified vessels
Variability of measurement | day 0-2 / day 4-10 / day 11-14
  For each patient, bilateal ultrasonography will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Clément GAKUBA, PhD, Principal Investigator — CHU CAEN
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
IPD won't be shared with other researchers. Data will be collected in a data base with an authentification by password. The used system is in accordance with the french law, notably MR-01. Only permitted person will be given an access to the data base. Every connection to the data base will be recorded.

REFERENCES:
- [Background] Ghendon Y. WHO recommendation on potential use of new poliomyelitis vaccines. Dev Biol Stand. 1993;78:133-7; discussion 138-9. PMID 8388823
- [Background] Shea SS, Selfridge-Thomas J. The ED nurse practitioner: pearls and pitfalls of role transition and development. J Emerg Nurs. 1997 Jun;23(3):235-7. doi: 10.1016/s0099-1767(97)90014-3. No abstract available. PMID 9283360
- See also: Clinical Application of Super-resolution Ultrasound(SR-US) Imaging in Solid Tumors — https://clinicaltrials.gov/study/NCT06018142
- See also: SUper-Resolution Ultrasound Imaging of Erythrocytes (SURE) in Normal and Malignant Lymph Nodes — https://clinicaltrials.gov/study/NCT05754814
- See also: Ultrasound Perfusion Imaging After Aneurysmal Subarachnoid Hemorrhage (PSAB) — https://clinicaltrials.gov/study/NCT01537263
- See also: Contrast Enhanced Ultrasound Imaging for Cerebral Perfusion Measurement in Cerebral Vasospasm After SAH — https://clinicaltrials.gov/study/NCT02907879